CLINICAL TRIAL: NCT00516867
Title: Sunbed Radiation Provoke Cutaneous Vitamin D Synthesis in Humans, a Randomized Controlled Trial
Brief Title: Does Sunbed Radiation With Mainly UVA Provoke Cutaneous Vitamin D Synthesis in Humans?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KF 01 290815
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ultraviolet Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- UVB 0.5% (Active Comparator)
  Interventions: Radiation: UV radiation
- Controls (No Intervention)
- UVB 1.4% (Active Comparator)
  Interventions: Radiation: UV radiation

INTERVENTIONS:
Radiation: UV radiation — UV radiation with 99.5% UVA and 0.5%UVB
  Arms: UVB 0.5%
Radiation: UV radiation — UVB 1.4 % and UVA 98.6
  Arms: UVB 1.4%

SUMMARY:
We would investigate in a controlled, randomized open study in the winter season: 1) If serum levels of vitamin D (25(OH)D) increase in subjects treated with sunbed with sunlamps emitting mainly UVA and only 0·5% or 1·4% UVB compared to non-sunbed treated controls 2) If yes, are the 25(OH)D serum levels then dependent on the UVB dose?

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Females
* Above 50 years
* Younger with serum concentration of 25(OH)D below 50nmol/l

Exclusion Criteria:

* No sunbed use last ½ year
* No sun holiday last ½ year
* No intake of vitamin D above 10 microgram/day

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-02; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Serum concentration of 25(OH)D | 18 Days

SECONDARY OUTCOMES:
Serum concentration of PTH | 18 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hans C Wulf, MD, DSc, Study Chair — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark